CLINICAL TRIAL: NCT04387032
Title: The Influence of the Sacroiliac Joint Manipulation on Changes in the Values of the Center of Pressure in the Process of Maintaining Static Body Balance
Brief Title: Impact of Manipulation of Sacroiliac Joints on the Static Balance of the Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Małgorzata Waszak, Study Director, Poznan University of Physical Education
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVLA manipulations
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Asymptomatic Condition; Sacroiliac Disorder
Keywords: manual therapy; HVLA manipulation; sacroiliac joint; center of pressure (COP); hypomobility
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Experimental group - HVLA manipulations on blocked sacroiliac joints (SIJs) Control group (people without hypomobile SIJs), in which we performed sham manipulation
Who Masked: Participant, Outcomes Assessor
Masking Description: blinded patient blinded researcher and person evaluating results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group (students with hypomobile SIJs)
  Interventions: Other: HVLA Manipulations
- Control group (Sham Comparator): control group (students without hypomobile SIJs)
  Interventions: Other: Sham Manipulation

INTERVENTIONS:
Other: HVLA Manipulations — The procedure of experimental manipulation: the patient lay on the healthy side with the straight lower limb, and the torso turned towards the dysfunctional side, whose lower limb was bent in the hip and knee joint, and the hands rest on the lower ribs on the same side. The therapist allowed the initial loosening of the tissues and chose the movement barrier with his stabilizing hand. Then, with the treatment hand, he introduced the HVLA thrust through the iliac bone towards the bottom, while giving the iliac bone a posterior or anterior rotation - meaning, the opposite to the occurring dysfunction. If during the manipulation, no cavitation sound was heard, the HVLA thrust was repeated once.
  Other Names: manual therapy
  Arms: Experimental group
Other: Sham Manipulation — The sham procedure was the same, but no external force was introduced in the form of a therapeutic impulse.
  Arms: Control group

SUMMARY:
The study can be identified as an experimental study with a quasi-randomized control. It consisted of HVLA manipulation on blocked sacroiliac joints (SIJ) and it was checked whether it affected the appropriate parameters determining the pressure center (COP). The value of the parameters were examined twice, before (PRE) and after (POST) manipulation. The results were compared with the control group (people without hypomobility SIJ) in which sham manipulation was performed, and COP parameters (PRE and POST) were measured twice. In addition, PRE and POST results were compared within the group, i.e. separately in the experimental group (E) and separately in the control group (C) to check the effect of HVLA manipulation and placebo manipulation.

The first hypothesis assumes that persons belonging to the experimental group are characterized by significantly higher values of COP parameters before manipulation than values in the control group. The second hypothesis assumes that COP parameters will normalize as a result of sacroiliac joint mobilization performed in the experimental group.

DETAILED DESCRIPTION:
The aim of the project was to determine the effectiveness of HVLA manipulation in maintaining static body balance. To implement it, it was necessary to conduct an experiment consisting in performing HVLA manipulation in people with SIJs hypomobility and checking whether it affects the COP parameters. It was assumed to measure these parameters twice (before (PRE) and after (POST) manipulation) and compare them with the measurements in the C group (sham manipulation).

The sample size necessary to power the study was determined at the test planning stage, using the G * Power 3.1.9 software. The standard threshold α = .05 was established; then the acceptable power level of the 1-β = .90 test and the expected moderate effect size η2 = .30 were determined for within-between interaction. The calculated total expected size of the sample is N = 32, i.e. 16 subjects in one research group, assuming that their number will not decrease during the study. With a higher test power 1-β = .95 and a moderate achieved result for observed effect size η2 = .25, the sample should have to consist of 26 subjects per subgroup. It was decided to examine a slightly larger number of available entities due to the possibility of excluding incorrect data.

Poznan University of Physical Education's students were invited to the research, electronically. Before starting the research, they were informed about the purpose and manner of conducting the research, and the type of methods used. Participation in the experiment was voluntary and free. Participants could withdraw from cooperation in the research at any time. They obtained assurance that the data obtained will be used only for scientific purposes and their processing will be fully anonymous.

Among 202 students of the Poznań University of Physical Education who responded to the invitation to the study project interview has been conducted, as a result of which 22 people were excluded from further actions due to disqualification criteria. Then sacroiliac mobility tests has been performed which made it possible to recognize hypomobility in 72 people. From the group of people with hypomobility, 36 people were randomly selected and included in the E group. From among people without hypomobility, 31 people were randomly selected for the C group. An random number table was used in the draw. The subjects did not know any group they were assigned to.

Subsequently, the examination of each project participant consisted of performing podometric measurements and SIJs mobilization in the E group or placebo in the C group, and re-performing functional tests and podometrics in both groups after the procedure. At the stage of analyzing data rejected 8 people who did not meet the assumed criteria, thus finally there were 30 people in the experimental group and 29 in the control group.

Functional tests

Qualification of the subjects to the E and C group was conducted by a researcher who had seven years of experience in using manual therapy techniques. The following tests of SIJs mobility were performed:

1. Standing forward flexion test: the symmetry of posterior superior iliac spine (PSIS) displacement during forward flexion is assessed. In the case of hamstrings tension, the result may be false positive, so it should be repeated in a sitting position or with slightly bent knees.
2. One leg standing / Stork / Gillet test: the hip joint is bent in the standing position, the downward and medial displacement of PSIS in relation to S2 is observed.
3. Measurement of the Derbolowsky symptom (Pidellou symptom / long sitting test): was performed as determined by Bemis and Daniel. It allows determining the dysfunctional side and the rotation of iliac bone. The level of medial ankles during lifting of the torso from lying back position to straight sit with simultaneous traction of legs is observed.
4. Lower limb adduction test: the patient is lying back, upper anterior iliac spine stabilization (ASIS) is required. The adduction of the bent at the hip and knee joint lower limb follows it. On the limited side, the adduction angle will be smaller compared to the healthy side. The test has screening character, because blockage of the joint may occur without limitation of adduction in the case of hip over-mobility, but due to the simplicity of implementation, it is a valuable indicator.

The majority of SIJs mobility tests are burdened with the accuracy and reliability errors in situations when they are performed individually. However, performing more tests increases the accuracy of the diagnosis. For this reason, there were performed four SIJs mobility tests, as well as complementary measurements of PSIS, ASIS, and iliac crest levels before (PRE) and after (POST) treatment to determine its effectiveness.

Podometric measurement After conducting functional tests, the study participants were directed to a podometric measurement, which was performed twice - PRE and POST. The measurement was carried out using the Medicapteurs PEL 38 platform, which allows conducting both static and dynamic measurements, and it cooperates with the TWINN software in Windows. The equipment was designed and tested in leading medical centers in Europe and put into use in the USA by Physical Support Systems. The platform has 1024 sensors with a total measuring surface of 320x320 [mm] and the appropriate resolution for testing the distribution of foot pressure and tracking the position of COP. The platform was calibrated automatically accordingly to the bodyweight of each participant, and the measurement was taken in a standing (Frankfurt) position with upper limbs hanging freely. Participants were asked to maintain a stable position without unnecessary movements and to look straight ahead at eye level. During the study, patients did not have visual access to a graphical record of the measurement carried out to avoid attempts to correct body posture. Each measurement was conducted for 30 seconds, recording the current COP position at a frequency of 10 frames per second.

Experimental manipulation Persons with blocked SIJ on one or both sides, constituting an E group, were manipulated on the blocked joints. People without blocked SIJs constituted a C group that underwent placebo manipulation.

The procedure of experimental manipulation: the patient lay on the healthy side with the straight lower limb, and the torso turned towards the dysfunctional side, whose lower limb was bent in the hip and knee joint, and the hands rest on the lower ribs on the same side. The therapist allowed the initial loosening of the tissues and chose the movement barrier with his stabilizing hand. Then, with the treatment hand, he introduced the HVLA thrust through the iliac bone towards the bottom, while giving the iliac bone a posterior or anterior rotation - meaning, the opposite to the occurring dysfunction. If during the manipulation, no cavitation sound was heard, the HVLA thrust was repeated once. In the C group, the placebo procedure was the same, but no external force was introduced in the form of a therapeutic impulse.

Statistical methods The collected data were analyzed in a statistical program Statistica version 13. The normality of the distribution of all measured variables on the quantitative scale in both groups was checked by the Shapiro-Wilk test .

In order to study the effect of the manipulation on the measured variables, there was carried out quantitative analysis of variance with repeated measures, plus a number of comparisons using the Student's t-test for dependent and independent attempts, and in some cases for the characteristics whose distribution differed from the standard - with the use of non-parametric the Mann-Whitney U-test for independent pairs or Wilcoxon test for dependent pairs. The Cohen d effect power measure was also used in data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Student at the Poznan University of Physical Education;
* age 19-24;
* asymptomaticity in the form of no pain symptoms in the LS segment of the spine;
* written consent to participate in the study;
* presenting no disqualification criteria;
* no health contraindications to perform manipulation;
* no hypomobility of the SI joints, negative mobility test results PRE (to the control group);
* occurrence of hypomobility of the SI joint on one or both sides PRE (to the experimental group);
* noting the sound of cavitation during the procedure (in the experimental group);
* confirmation of a treatment effectiveness by noting negative results of SI joints mobility tests POST (in the experimental group).

Exclusion Criteria:

Persons who were characterized by LBP, neurological symptoms, rheumatic problems, orthopedic, or ongoing treatment in the lumbar spine and pelvis area were excluded. Pregnancy and the anatomical difference in the length of the lower limbs exceeding 5mm were also an excluding criterion.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
COP X PRE | PRE (immediately before the intervention)
  deflection of the COP in the X axis before manipulation
COP X POST | POST (immediately after the intervention)
  deflection of the COP in the X axis after manipulation
COP Y PRE | PRE (immediately before the intervention)
  deflection of the COP in the Y axis before manipulation
COP Y POST | POST (immediately after the intervention)
  deflection of the COP in the Y axis after manipulation
COP Length PRE | PRE (immediately before the intervention)
  path travelled by COP before manipulation;
COP Length POST | POSt (immediately after the intervention)
  path travelled by COP after manipulation;
COP Area PRE | PRE (immediately before the intervention)
  COP area before manipulation
COP Area POST | POST (immediately after the intervention)
  COP area after manipulation
COP Av.Q-speed PRE | PRE (immediately before the intervention)
  the average speed of COP before manipulation
COP Av.Q-speed POST | POST (immediately after the intervention)
  the average speed of COP after manipulation

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Waszak, PhD, Study Director — Poznan University of Physical Education; Michał Posłuszny, MSc, Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Department of Biology and Anatomy, Poznan, Wielkopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
University IPD sharing platform is under preparation. All data will also be available to researchers via the study's director email (waszak@awf.poznan.pl) or Research Gate website.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from June 2020.
Access Criteria: Available to all researchers
URL: http://www.awf.poznan.pl/pl/noz-anatomia-biologia-aktualnosci

REFERENCES:
- [Background] Vleeming A, Schuenke MD, Masi AT, Carreiro JE, Danneels L, Willard FH. The sacroiliac joint: an overview of its anatomy, function and potential clinical implications. J Anat. 2012 Dec;221(6):537-67. doi: 10.1111/j.1469-7580.2012.01564.x. Epub 2012 Sep 19. PMID 22994881
- [Background] Coulter ID, Crawford C, Hurwitz EL, Vernon H, Khorsan R, Suttorp Booth M, Herman PM. Manipulation and mobilization for treating chronic low back pain: a systematic review and meta-analysis. Spine J. 2018 May;18(5):866-879. doi: 10.1016/j.spinee.2018.01.013. Epub 2018 Jan 31. PMID 29371112
- [Background] Lord SR, Clark RD, Webster IW. Physiological factors associated with falls in an elderly population. J Am Geriatr Soc. 1991 Dec;39(12):1194-200. doi: 10.1111/j.1532-5415.1991.tb03574.x. PMID 1960365
- [Background] Bemis T, Daniel M. Validation of the Long Sitting Test on Subjects with lliosacral Dysfunction*. J Orthop Sports Phys Ther. 1987;8(7):336-45. doi: 10.2519/jospt.1987.8.7.336. PMID 18797042
- [Background] Arab AM, Abdollahi I, Joghataei MT, Golafshani Z, Kazemnejad A. Inter- and intra-examiner reliability of single and composites of selected motion palpation and pain provocation tests for sacroiliac joint. Man Ther. 2009 Apr;14(2):213-21. doi: 10.1016/j.math.2008.02.004. Epub 2008 Mar 25. PMID 18373938
- [Result] Grassi Dde O, de Souza MZ, Ferrareto SB, Montebelo MI, Guirro EC. Immediate and lasting improvements in weight distribution seen in baropodometry following a high-velocity, low-amplitude thrust manipulation of the sacroiliac joint. Man Ther. 2011 Oct;16(5):495-500. doi: 10.1016/j.math.2011.04.003. Epub 2011 May 14. PMID 21570892
- [Result] Koes BW, Assendelft WJ, van der Heijden GJ, Bouter LM. Spinal manipulation for low back pain. An updated systematic review of randomized clinical trials. Spine (Phila Pa 1976). 1996 Dec 15;21(24):2860-71; discussion 2872-3. doi: 10.1097/00007632-199612150-00013. PMID 9112710
- [Result] von Heymann WJ, Schloemer P, Timm J, Muehlbauer B. Spinal high-velocity low amplitude manipulation in acute nonspecific low back pain: a double-blinded randomized controlled trial in comparison with diclofenac and placebo. Spine (Phila Pa 1976). 2013 Apr 1;38(7):540-8. doi: 10.1097/BRS.0b013e318275d09c. PMID 23026869
- [Result] Farazdaghi MR, Motealleh A, Abtahi F, Panjan A, Sarabon N, Ghaffarinejad F. Effect of sacroiliac manipulation on postural sway in quiet standing: a randomized controlled trial. Braz J Phys Ther. 2018 Mar-Apr;22(2):120-126. doi: 10.1016/j.bjpt.2017.09.002. Epub 2017 Sep 8. PMID 28993042